CLINICAL TRIAL: NCT06074107
Title: An Open, Multicenter Phase II Study of the Efficacy and Safety of BEBT-908 in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Study of BEBT-908 in the Relapsed or Refractory Diffuse Large B-cell Lymphoma Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-908-P02
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Relapsed or Refractory Diffuse Large B-cell Lymphoma
Keywords: BEBT-908; safety; efficacy
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — BEBT-908; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BEBT-908 for injection (Experimental): BEBT-908 for injection, dosage form: injection, specification: 25mg, administration method: the initial dose was 22.5mg/m2, intravenous drip, 3 times a week, 21 days as a cycle, 6 cycles as the total treatment cycle.
  Interventions: Drug: BEBT-908 for injection

INTERVENTIONS:
Drug: BEBT-908 for injection — The initial dose is 22.5mg/m2, intravenous drip, on the 1st, 3rd, 5th, 8th, 10th and 12th day of each cycle，21 days as a cycle, 6 cycles as the total treatment cycle.
  Other Names: CUDC-908

SUMMARY:
This is an open,single-arm,multicenter phase II clinical study to evaluate the efficacy and safety of BEBT-908 for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma. The study will be divided into two stages: phase Ⅱa and phase Ⅱb. Phase Ⅱa is an exploratory study, which mainly explores the safe and effective dose and the relationship between gene and protein markers and drug sensitivity. The main purpose of the phase Ⅱb study was to evaluate the Objective response rate of BEBT-908 for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma, and the secondary study was to evaluate the disease control rate, progression-free survival, time to response, duration of response, overall survival and safety tolerance of BEBT-908 for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma. The relationship between the biomarkers of BEBT-908 for injection and the efficacy and safety was evaluated.

DETAILED DESCRIPTION:
This is an open, single-arm, multicenter phase II clinical study to evaluate the efficacy and safety of BEBT-908 for injection in the treatment of relapsed or refractory diffuse large B-cell lymphoma. The study will be divided into two stages: Ⅱa and Ⅱb, stage Ⅱa is an exploratory study, which mainly explores the safe and effective dose, 30 cases are planned to be included in the group, stage Ⅱb mainly evaluates the efficacy and safety of BEBT-908 for injection, according to the preliminary overall efficacy analysis of stage Ⅱa, the sample size of stage Ⅱb is about 90 cases.

In phase Ⅱa and Ⅱb study, the initial dose was 22.5mg/m2, intravenous drip, 21 days as a cycle and 6 cycles as the total treatment cycle. The drugs were given on the 1st, 3rd, 5th, 8th, 10th and 12th day of each cycle. The study process of each subject included three periods: screening period, treatment period and follow-up period after treatment. During the treatment period, all safety items were examined before administration on the first day of each cycle, and the tumor was evaluated every 2 cycles. After the termination of treatment, the subjects will enter the follow-up period. Receive curative effect follow-up every 6 weeks (to tumor progression or other anti-tumor therapy) and survival follow-up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing to sign the informed consent form (ICF) after a comprehensive understanding.
2. Age ≥ 18 years and ≤ 75 years, male or female.
3. Diffuse large B-cell lymphoma was confirmed by central pathological examination and tissue biopsy.(Note 1)
4. With measurable lesions.(Note 2)
5. Refractory or relapse after at least two kinds of systematic treatment. (Note 3)
6. Eastern Cooperative Oncology Group (ECOG) score ≤ 2.
7. Life expectancy > 12 weeks.
8. The level of organ function must meet the following requirements:

Peripheral blood:

1. Absolute neutrophil count (ANC) ≥ 1000 /μL.
2. Hemoglobin (HGB) ≥ 8g/dL.
3. Platelet count (PLT) ≥ 1000000 /μL.

Liver function:

1. Serum total bilirubin ≤ 1.5 × Upper limit of normal value （ULN） (for patients with Gilbert syndrome, total bilirubin < 3.0 × ULN and direct bilirubin within the normal range).
2. Serum creatinine < 1.5 × ULN.
3. Alanine aminotransferase （ALT）, aspartate aminotransferase （AST） or alkaline phosphatase （ALP ）≤ 2.5 × ULN (≤ 5 × ULN when liver involvement is involved).

Note 1: Patients with recurrence for more than one year need to undergo another tissue biopsy to confirm the pathological diagnosis.

Note 2: the criteria for measurable lesions are as follows: the longest diameter of lymph node lesions is more than 15 mm under enhanced Computed Tomography （ （CT ）or Magnetic Resonance Imaging (MRI), the longest diameter of extranodal lesions is more than 10 mm, or the longest diameter of extranodal lesions is ≥ 10 mm under Positron Emission Tomography/Computed Tomography (PET/CT). Bone marrow aspiration cytology and / or biopsy may be performed when evaluating the curative effect.

Note 3: Relapsed / refractory diffuse large B lymphoma is defined in this regimen as: 1) relapsed more than 6 months after the end of second-line treatment; 2) those who relapse within 6 months after the end of second-line treatment and those who do not reach partial response (PR) for 2 or more cycles of second-line treatment can be selected as refractory patients without the requirement of treatment cycle. 3) after sequential hematopoietic stem cell transplantation with second-line therapy, recurrence within 6 months can be included in the group. Previous treatment should include anti-CD20 monoclonal antibody and cytotoxic drug therapy; anti-CD20 monoclonal antibody consolidation therapy or induction therapy cannot be counted as a single line of treatment; previous stem cell transplantation is allowed; autologous stem cell transplantation or allogeneic stem cell transplantation alone does not count as first-line therapy, induction, consolidation, stem cell collection, pretreatment regimen and transplantation ±maintenance therapy belong to the same line of treatment.

Exclusion Criteria:

1. It is known to be severely allergic to research drugs or any of their excipients.
2. Because the research drugs may have genotoxicity, mutagenicity and teratogenicity, the following subjects should be excluded:

   1. Men and women who plan to reproduce within 5 years without in vitro preservation of sperm or eggs before the trial. Unless follow-up studies confirm reproductive safety.
   2. pregnant or lactating women.
3. Primary central nervous system lymphoma or lymphoma invading the central nervous system.
4. Previous transformation of chronic lymphoma (such as Richter syndrome, pre-lymphocytic leukemia, etc.).
5. There are other active malignant tumors that may interfere with this study.
6. Pre-trial treatment:

   1. Have received any persistent or intermittent treatment such as Phosphoinositide 3-kinase (PI3K) inhibitors, Mammalian Target of Rapamycin (mTOR) inhibitors or Histone Deacetylase (HDAC) inhibitors or other small molecule targeted drugs within 2 weeks before entering the group.
   2. Autologous hematopoietic stem cell transplantation within 3 months before enrollment.
   3. Received radiotherapy that affected the efficacy evaluation of this study or local supportive radiotherapy that affected the bone marrow function of the subjects within 3 months before enrollment.
   4. Bone marrow inhibitory chemotherapy or biotherapy was performed within 3 weeks before enrollment.
   5. Major surgery other than tumor biopsy was performed within 4 weeks before enrollment, or the side effects of the operation were not stable.
   6. Received any hematopoietic colony-stimulating factor therapy (such as granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF)) or thrombopoietin （TPO） within 2 weeks before enrollment. (Note 1)
   7. received prednisone daily > 10mg (or other dose-effective corticosteroids) within 7 days before enrollment. (Note 2)
   8. Chimeric antigen receptor T cell immunotherapy (CAR-T therapy) was performed within 3 months before enrollment.
7. After the previous treatment (chemotherapy or biotherapy), there were persistent toxicity of grade 2 or above (Common Terminology Criteria for Adverse Events V5.0 （CTCAE V5.0 ）), which was not stable at the time of admission (except hair loss).
8. There are severe clinical infections in active stage with grade 2 or above (CTCAE V5.0).
9. Concomitant disease:

   1. Diabetes with poor blood glucose control (random blood glucose ≥ 11.1mmol/L or Hemoglobin A1C (HbA1c ）≥ 8.5% after hypoglycemic treatment).
   2. Severe lung disease (CTCAE V5.0, III-IV).
   3. Severe heart disease. (Note 3)
   4. With significant renal or liver dysfunction.
   5. Poorly controlled active hepatitis B or C diseases;(Note 4)
   6. known to be HIV positive.
   7. A history of mental illness, family history of mental illness or emotional disorder is determined by a researcher or psychiatrist. (Note 5)
10. Combined use of drugs that cause prolonged QT interval or twisted ventricular tachycardia.
11. The patients were treated with cytochrome P450 (CYP) 3A4 isozyme inhibitors or strong induction drugs within 4 weeks before enrollment. (Note 6)
12. Participated in other clinical trials and used research drugs within 4 weeks before joining the group.
13. The researchers judged any unstable or likely to endanger the safety of subjects and their compliance with the study.
14. The researchers believe that it is not suitable for subjects who are treated with this regimen.

Note 1: Subjects who began to receive erythropoietin or diplotene within 2 weeks before enrollment can be enrolled in the group.

Note 2: If used to treat diseases other than lymphoma, such as rheumatoid arthritis, rheumatic polymyalgia, adrenocortical dysfunction or asthma, subjects can receive a maximum daily dose of 10mg with a stable dose of prednisone (or other equivalent glucocorticoid).

Note 3: Including any of the following: left ventricular ejection fraction (LVEF) < 50% found by cardiac radionuclide scanning (Multigated Radionuclide Angiography （MUGA）) or echocardiography (ECHO) corrected QT value (QTcF interval) male > 450ms, female > 470ms (QTcF formula); unstable angina pectoris; symptomatic pericarditis; abnormal recording of the left ventricular wall in areas with persistent elevated myocardial enzymes or persistent LVEF function measurements in the past 6 months of myocardial infarction.

History of congestive heart failure (New York College of Cardiology III-IV Appendix 3), cardiomyopathy record.

Note 4: The following active infections with clinical significance, including hepatitis B (HBV) and hepatitis C (HCV). Active hepatitis B is defined as hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg) positive, and HBV DNA ≥ 2000 IU/ml (equivalent to 10^4 copies / ml), (hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg) positive, HBV DNA < 2000 IU/ml, according to infectious disease control requirements, subjects should continue to take entecavir until one year after the end of the study). Active hepatitis C is defined as: HCV RNA is higher than the upper limit of detection.

Note 5: including medical records with history of depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, suicidal attempts or suicidal ideations, or thoughts of "being at immediate risk of harming others", anxiety level 3 or above, etc.

Note 6: moderate or weak CYP3A inhibitors are allowed in combination; a list of common CYP3A4 inhibitors or inducers is shown in Appendix 5 of the study scheme.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 weeks， assessed up to 24 months.
  Objective response rate

SECONDARY OUTCOMES:
DCR | Every 6 weeks， assessed up to 24 months.
  Disease Control Rate
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Progress Free Survival
TTR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Time to Response
DOR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Duration of Response
OS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Overall Survival
AE | From the first administration of the study drug to 30 days after the last administration of the study drug.
  Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Phd, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China